CLINICAL TRIAL: NCT06814405
Title: Safety and Feasibility of a Multidisciplinary Programme of Integrated Hospital-home Management With Early Discharge of Patients With Haematological Malignancies Undergoing High-dose Chemotherapy in Hospital
Acronym: AMICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMICO; AIL Bologna (Other Grant/Funding Number: AIL Bologna ODV)
Record Dates: First submitted 2024-12-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Haematological Malignancy
Keywords: hospitalisation; early discharge; domiciliation; supportive therapy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hospitalized (Active Comparator): Hospedalized patients
  Interventions: Other: Hospital patient management
- early discarged (Experimental): Early discarged patients
  Interventions: Procedure: Home patient management

INTERVENTIONS:
Procedure: Home patient management — with support therapy, Granulocyte growth factor, blood transfusion
  Arms: early discarged
Other: Hospital patient management — all procedures and exams needed
  Arms: hospitalized

SUMMARY:
Patients undergoing particular intensive and (sub)myeloablative chemotherapy regimens with subsequent autologous stem cell transplant currently have a relatively low rate of therapy-related complications, both infectious and non-infectious (organ damage), and can therefore benefit from a specific multidisciplinary care programme at home. In this clinical context, early discharge and domicile of the patient after therapy provided in a hospital setting may represent a procedure designed to better intercept the patient's personal needs. In addition, it may make it possible to increase the limited availability of beds in the face of the progressive increase in demand, allowing the provision of hospital therapies to a higher number of patients with a consequent reduction in pre-hospital waiting times.

DETAILED DESCRIPTION:
Patients undergoing particular intensive and (sub)myeloablative chemotherapy regimes with subsequent autologous stem cell transplant currently have a relatively modest rate of therapy-related complications, of infectious and non-infectious (organ damage), relatively modest, thus being able to benefit of a specific multidisciplinary care programme at home. In this clinical context, the early discharge and domicile of the patient after therapy provided in hospital regimen may represent a procedure designed to better intercept the patient's patient's personal needs. In addition, it may make it possible to increase the limited availability of beds against the progressive increase in demand, allowing the provision of hospital treatment to a higher number of patients with a consequent reduction in pre-admission waiting times. The primary objective of the study is to assess the safety and feasibility of the model of early discharge with home continuation of the care pathway of patients haematological patients undergoing high-dose chemotherapy with/without autologous stem cell transplant.

The secondary objectives are as follows:

* Assessment of the patient's quality of life;
* Evaluation of the impact of the use of innovative remote monitoring technologies;
* Assessment of the optimisation of in-patient places;
* Evaluation of the economic impact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of haematological malignancy undergoing high-dose chemotherapy (sub- or myeloablative)
* Age between 18-75 years
* WHO Performance Status < 2 or Karnofsky ≥ 60%
* Adequate organ function:
* FE≥ 50% and absence of significant electrocardiographic changes
* eVFG > 40 ml/min and/or creatinine ≤ 1.6 mg/dl (CPK-EPI formula)
* total bilirubin ≤ 3 mg/ml
* AST/ALT ≤ 5 ULN
* SpO2 ≥ 94%
* Reinfusion ≥ 2x106 CD34+/Kg
* Presence of a 24-hour SARS-COV-2 vaccinated caregiver
* Home < 45 minutes' drive from hospital
* Informed consent obtained

Exclusion Criteria:

* Diagnosis of haematological malignancy at onset or in progression
* Significant cardiovascular disease: heart failure NYHA class 3 or 4, uncontrolled angina, history of myocardial infarction, unstable angina or stroke in the previous 6 months, uncontrolled hypertension, significant arrhythmias not controlled by medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | through the duration of study, an average of 2 years
  safety of the early discharge model with home continuation of the care pathway of haematological patients undergoing high-dose chemotherapy with/without autologous stem cell transplant
Number of participants in which will be feasible the early discarge mode | through the duration of study, an average of 2 years
  feasibility of the early discharge model with home continuation of the care pathway of haematological patients undergoing high-dose chemotherapy with/without autologous stem cell transplant

SECONDARY OUTCOMES:
questionnaire patient's quality of life FACT-An (Functional Assessment of Cancer Therapy) (V. 4, scale 0-4) | through the duration of study, an average of 2 years
  Assessment of the patient's quality of life with questionnaire FACT-An(Functional Assessment of Cancer Therapy) (V. 4, scale 0-4) at early discharge and recovery hematology
Median length of stay with early discharge (outpatient)/median length of hospitalization without early discharge (inpatient) of patients who were enrolled but, for reasons various, were not discharged early; | through the duration of study, an average of 2 years
  Median length of stay with early discharge (outpatient)/median length of hospitalization without early discharge (inpatient) of patients who were enrolled but, for reasons various, were not discharged early;
rate of optimisation of in-patient places | through the duration of study, an average of 2 years
  Assessment of optimisation of in-patient places
Rate of Economic Impact | through the duration of study, an average of 2 years
  Economic Impact Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS-AOU di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No